CLINICAL TRIAL: NCT02552901
Title: A Pivotal, Within Subject, Comparison of the LFT™ Dye Monitor System to the Indocyanine Green Dye (ICG) Serial Blood Plasma Disappearance Rate in Patients With Impaired and Non-Impaired Hepatic Function
Brief Title: Cardiox Liver Function Test Pivotal Trial
Acronym: LFT-0002
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LFT-0002
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Failure; Liver Failure
Keywords: hepatic; liver; LFT; hepatic assessment; ICG dye; indocyanine green dye; Diagnostic Green; Pulsion; Akorn; Cardiox; anazen; essence; dye detection monitor; Earpads; flow sensor; scaphoid fossa; liver disease; acute hepatic failure; AHF; NASH; hepatitis C; cirrhosis; MELD; pulse dye densitometry; liver transplant; fluorescence; near infra-red; serial blood draws; PDR; plasma disappearance rate; R15; k coefficient; transcutaneously; liver donor; liver dysfunction; Child-Pugh; AST; ALT; GGT; alk phos; prothrombin time; albumin; serum ICG; liver function tests
MeSH Terms: conditions — Liver Failure; Liver Diseases; Liver Failure, Acute; Hepatitis C; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LFT Dye Detection Monitor (Experimental)
  Interventions: Drug: 0.1 mg/kg ICG Dose; Drug: 0.5 mg/kg ICG dose
- Serial Blood Draws (Active Comparator)
  Interventions: Drug: 0.5 mg/kg ICG dose

INTERVENTIONS:
Drug: 0.1 mg/kg ICG Dose — least efficacious dose
  Other Names: LFT Dose
  Arms: LFT Dye Detection Monitor
Drug: 0.5 mg/kg ICG dose — per package insert

SUMMARY:
Performance evaluation of LFT Dye Monitor System using ICG - plasma disappearance rate value (PDR) to assess liver function in normal patients as well as in patients with mild to severe hepatic impairment compared to manual Serum ICG PDR.

DETAILED DESCRIPTION:
Indocyanine green (ICG) is a water-soluble, non-toxic tricarbocyanine dye, extracted principally by hepatic parenchymal cells and excreted almost entirely into the bile without enterohepatic circulation. Clinically, its elimination rate is used primarily to measure hepatic function and liver blood flow. ICG studies are also used in ophthalmic angiography and the determination of cardiac output.

Beginning about 1959, the first human clinical studies were reported wherein an indocyanine green (ICG) bolus was injected into a vein, and then blood samples were withdrawn over a period of time and analyzed for ICG concentrations. This method is referred to hereinafter as the serial blood sampling method. These blood samples are sent to a clinical laboratory for a multi-step process of centrifuging, separation and spectrophotometric measurements of ICG levels. The laboratory-based measured levels of residual ICG levels are then used to determine the ICG clearance rate and R15 value or residual amount of dye remaining after 15 minutes, expressed as a percentage of the initial concentration.

As an alternative to the time- and labor-consuming serial blood sampling method, a non-invasive technique was first reported nearly 20 years ago. In the first published clinical study, Ishigami reported the use of a pulse dye densitometry (PDD) method to transcutaneously detect the rate of clearance of ICG from the bloodstream to be referred to hereinafter as dynamic liver function testing.

PDD expresses ICG elimination in terms of the indocyanine green plasma disappearance rate because only relative ICG concentration changes are assessed. The results of this noninvasive method have been shown to correlate with those obtained by the invasive method used in critically ill patients (hemodynamically unstable and stable), and in patients after liver surgery.

ICG elimination rate after liver transplantation measured by either invasive or noninvasive ICG methods is widely used to evaluate graft function. Studies have shown that ICG elimination, measured on the day of transplantation, reflects graft function and can be used to predict graft viability and the expected survival of the patient. Sequential measurements of ICG elimination between days 0 and 28 of transplantation, have been shown to predict clinical outcome in the early postoperative period after living donor transplantation. All of the studies have shown that the ICG elimination rate is an accurate test for evaluating liver dysfunction, but lacks the ability to differentiate the underlying causes of the hepatic dysfunction.

Unlike all currently existing PDD methods for performing liver function testing, LFT Dye Monitor System employs a more sensitive method for the transcutaneous measurement of ICG concentration level in the blood using NIR fluorescence, with a sensor that is attached loosely to the scaphoid fossa of the ear. Thus, the chemical properties of ICG dye to fluoresce when properly excited are used in the LFT system to enable much lower concentrations of ICG to be detectable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 to 75 years of age inclusive, at the time of Screening.
2. Voluntarily provide written informed consent.
3. Female patients are eligible only if all of the following apply:

   * Not pregnant (negative urine pregnancy test at the Screening visit);
   * Not lactating;
   * Not planning to become pregnant within the duration of the study;
   * Surgically sterile, or at least 2 years postmenopausal, or is practicing an acceptable form of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, subdermal implant, oral contraceptives, abstinence, or sterilization of monogamous partner) for greater than 60 days prior to Screening and commits to the use of the acceptable form of birth control for the duration of the study.
4. If a healthy volunteer; is considered to be in generally good health, in the opinion of the Investigator, at the Screening visit based upon the results of their medical and surgical history, vital signs, physical examination, and clinical laboratory tests.
5. Prior to receiving any ICG injections the subject agrees to be fasting for at least eight (8) hours.
6. If a subject with liver cirrhosis; is considered to be in general satisfactory health, in the opinion of the Investigator (other than their hepatic impairment) at the Screening visit based upon the results of their medical and surgical history, vital signs, physical examination, and non-hepatic clinical laboratory tests.
7. Liver cirrhosis subjects must have a clinical diagnosis of hepatic impairment based on documented evidence of hepatic cirrhosis by medical history, or previous liver biopsy, or hepatic ultrasound; which conforms to the criteria for class A or B or C of the Childs-Pugh classification (Appendix B); and are expected to require an ICG liver function study, such as for liver transplantation, liver resection, liver cirrhosis prognosis evaluation, functional liver cell mass and/or general liver dysfunction evaluations.
8. On stable drug therapy that is not expected to change (i.e. in dose, frequency, additions or deletions of agents) for at least 2 weeks before ICG dye injection.
9. Must, in the Investigator's opinion, be able to comply with study procedures.
10. If the Subject is being enrolled in the fifth group they have a diagnosis of acute liver failure (ALF) as defined by the Principal Investigator.

Exclusion Criteria:

1. Have any clinically significant condition or unstable current illness that would, in the opinion of the Investigator, preclude study participation or interfere with the assessment of the procedure;
2. Known allergy or sensitivity to ICG dye or history of allergy to iodides;
3. Actively bleeding associated with acute blood volume changes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
plasma disappearance rate | Study Day 1

SECONDARY OUTCOMES:
physical examinations | Study Day 1
vital signs | Study Day 1
adverse events | Study Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jopling, MD, Study Director — Medical Director, Cardiox Corporation
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States